CLINICAL TRIAL: NCT07363993
Title: Interaction Between Intraventricular Flow and Cardiac Mechanics Using 3D Echocardiography in Athletes and Sedentary Subjects
Acronym: CARDIO-3D
Status: Recruiting | Type: Observational
Sponsor: University of Avignon (Other)
Collaborators: CHU Arnaud de Villeneuve MONTPELLIER (Unknown)
Responsible Party: Sponsor
Other Study IDs: AU-112025-CM; LAPEC/2025/CARDIO-3D (Other: Avignon University)
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Athlete Heart
Keywords: regional myocardial function; intraventricular flow; cardiac geometry; echo-3D; athlete's heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Sedentary controls
- Athletes: Endurance athletes

SUMMARY:
Exercise-induced cardiac remodeling, known as the "athlete's heart," corresponds to morphological and functional adaptations of the left ventricle in response to prolonged physical training. It is characterized in particular by physiological hypertrophy and improved myocardial function.

Intraventricular blood flow interacts with cardiac mechanics. Regional shape (e.g., sphericity, wall curvature) and myocardial deformations guide flow patterns to create an optimal hemodynamic environment. The interaction between these different parameters in the athlete's heart remains insufficiently explored. In this context, 3D echocardiography makes it possible to combine indices derived from fluid dynamics, regional myocardial function, and cardiac geometry, enabling a comprehensive assessment of cardiac performance.

Primary and secondary objectives:

In this context, the aim of this project is to investigate the relationship between intraventricular flow and cardiac mechanics based on combined measurements of intraventricular flow (e.g., vorticity, pressure gradients), regional myocardial function (e.g., myocardial strain), and global/regional LV geometry (e.g., sphericity, wall curvature) in the athlete's heart. Since these parameters are interdependent, analyzing their interaction through the development of new echocardiographic tools based on 4D assessments will enable a comprehensive evaluation of functional improvements in the athlete's heart.

The secondary objectives are to analyze the impact of dyssynchrony on intraventricular flow, to evaluate the influence of primary and secondary deformations on intraventricular flow, and to study cardiac function from an energetic perspective using non-invasive reconstruction of pressure-volume loops for cardiac work estimation.

Methodology:

The study will include 80 endurance athletes (ENT group) and 80 control subjects (CONT group). The main inclusion criteria common to both groups are: men and women aged 18-45 years, with no known heart disease and no cardiovascular risk factors (e.g., body mass index > 30 kg/m², arterial hypertension). Athletes must train at least 10 hours per week for the past 5 years. Control subjects must not engage in more than 3 hours of physical activity per week.

Athletes will be recruited from elite groups of various federations, during local long-distance races, or during clinical evaluations at Montpellier University Hospital (Dr. C. Hédon's department). Control subjects will be recruited in the Avignon area and in the cardiology department of Montpellier University Hospital during routine visits.

Echocardiographic examinations will be performed in the left lateral decubitus position using Vivid systems with 4D probes. 4D and tri-plane acquisitions with color Doppler will allow assessment of cardiac structure and intraventricular flow. Data analysis will be performed using TOMTEC software, and scripts developed in Matlab and RStudio will process information related to shape, mechanical dispersion, and dyssynchrony. Intraventricular hemodynamics will be analyzed in collaboration with the CREATIS laboratory (D. Garcia), particularly through measurements of intraventricular pressure gradients and vorticity indices.

ELIGIBILITY:
Inclusion criteria for athletes:

- Athlete practicing at least 10 hours of endurance training per week for a minimum of 5 years.

Inclusion criteria for controls:

- Individual not training in more than 3 hours of physical activity per week.

Exclusion Criteria for both groups:

* History of known heart disease;
* Current cardiac rhythm disorder;
* Individual with one or more cardiovascular risk factors (smoking, diabetes, hypertension, body mass index > 30 kg/m²);
* Individual in a period of relative exclusion in relation to another protocol, or for whom the annual maximum compensation amount of €4,500 has been reached;
* Individual not affiliated with a social security system, or not benefiting from such a system;
* Pregnant or breastfeeding woman; patient unable to give informed consent; protected adults; vulnerable persons;
* Individual deprived of liberty by judicial or administrative decision.

Exclusion criteria for athletes:

- Use of substances listed on the prohibited substances list of the French Anti-Doping Agency

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in the ENT group will be recruited:
  * At Montpellier University Hospital, in the cardiology department of Dr Hédon, during a follow-up visit.
  * At various national training centers of the French Triathlon Federation and the French Athletics Federation;
  * During local long-distance events (e.g., long-distance triathlons, ultramarathons), with assessments carried out at the time of race bib collection.
  Healthy participants will be recruited in parallel In Avignon and the surrounding area.
  Some participants from the CONT or ENT groups will also be recruited in the cardiology department of Dr Hédon at Montpellier University Hospital during a follow-up visit, for example as part of systematic cardiovascular screening. These participants will have undergone a preventive cardiology consultation that revealed no abnormalities or pathology. If these participants meet all inclusion criteria, they may then be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular principal strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular principal strains in resting conditions using 3D echocardiography in the two groups.

SECONDARY OUTCOMES:
Left ventricular secondary strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular secondary strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular principal and secondary strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular principal and secondary strain rates in resting conditions using 3D echocardiography in the two groups.
Left ventricular global longitudinal strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global longitudinal strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular global longitudinal strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global longitudinal strain rates in resting conditions using 3D echocardiography in the two groups.
Left ventricular global circumferential strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global circumferential strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular global circumferential strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global circumferential strain rates in resting conditions using 3D echocardiography in the two groups.
Left ventricular global radial strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global radial strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular global radial strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global radial strain rates in resting conditions using 3D echocardiography in the two groups.
Left ventricular global area strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global area strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular global area strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global area strain rates in resting conditions using 3D echocardiography in the two groups.
Standard deviation of the time-to-peak of left ventricular segmental strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess standard deviation of the time-to-peak of left ventricular segmental strains in resting conditions using 3D echocardiography in the two groups.
Maximum delay | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess maximum delay of left ventricular segmentary strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular longitudinal strain delay index | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular longitudinal strain delay index in resting conditions using 3D echocardiography in the two groups.
Left ventricular post systolic strain index | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular post systolic strain index in resting conditions using 3D echocardiography in the two groups.
Left ventricular myocardic work | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will left ventricular myocardic work in resting conditions using 3D echocardiography in the two groups.
Left ventricular potential energy | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular potential energy in resting conditions using 3D echocardiography in the two groups.
Right ventricular global longitudinal strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular global longitudinal strains in resting conditions using 3D echocardiography in the two groups.
Right ventricular global longitudinal strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular global longitudinal strain rates in resting conditions using 3D echocardiography in the two groups.
Right ventricular global circumferential strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular global circumferential strains in resting conditions using 3D echocardiography in the two groups.
Right ventricular global circumferential strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular global circumferential strain rates in resting conditions using 3D echocardiography in the two groups.
Right ventricular principal strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular principal strains in resting conditions using 3D echocardiography in the two groups.
Right ventricular secondary strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular secondary strains in resting conditions using 3D echocardiography in the two groups.
Right ventricular principal strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular principal strain rates in resting conditions using 3D echocardiography in the two groups.
Right ventricular secondary strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular secondary strain rates in resting conditions using 3D echocardiography in the two groups.
Right ventricular global area strain | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular global area strains in resting conditions using 3D echocardiography in the two groups.
Right ventricular global area strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular global area strain rates in resting conditions using 3D echocardiography in the two groups.
Left atrial global longitudinal strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left atrial global longitudinal strains in resting conditions using 3D echocardiography in the two groups.
Left atrial global longitudinal strain rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left atrial global longitudinal strain rates in resting conditions using 3D echocardiography in the two groups.
Right atrial global longitudinal strains | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right atrial global longitudinal strains in resting conditions using 3D echocardiography in the two groups.
Left ventricular global longitudinal strains - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global longitudinal strains in resting conditions using 2D echocardiography in the two groups.
Left ventricular global longitudinal strain rates - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global longitudinal strain rates in resting conditions using 2D echocardiography in the two groups.
Basal rotation - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular basal rotation in resting conditions using 2D echocardiography in the two groups.
Apical rotation - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular apical rotation in resting conditions using 2D echocardiography in the two groups.
Basal rotation - 3D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular basal rotation in resting conditions using 3D echocardiography in the two groups.
Apical rotation - 3D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular apical rotation in resting conditions using 3D echocardiography in the two groups.
Left ventricular twist | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular twist in resting conditions using 2D echocardiography in the two groups.
Left ventricular torsion | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular torsion in resting conditions using 3D echocardiography in the two groups.
Left ventricular twisting/untwisting rates - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular twisting/untwisting rates in resting conditions using 2D echocardiography in the two groups.
Left ventricular torsional rates - 3D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular torsional rates in resting conditions using 3D echocardiography in the two groups.
Left ventricular basal/apical rotational rates | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular basal/apical rotational rates in resting conditions using 2D echocardiography in the two groups.
Left ventricular circumferential strains - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess regional left ventricular circumferential strains in resting conditions using 2D echocardiography in the two groups.
Left ventricular circumferential strain rates - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular regional circumferential strain rates in resting conditions using 2D echocardiography in the two groups.
Left ventricular global myocardial work - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular global myocardial work in resting conditions using 2D echocardiography in the two groups.
Left ventricular myocardial constructive work - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular myocardial constructive work in resting conditions using 2D echocardiography in the two groups.
Left ventricular myocardial wasted work - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular myocardial wasted work in resting conditions using 2D echocardiography in the two groups.
Left ventricular myocardial work efficiency - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular myocardial work efficiency in resting conditions using 2D echocardiography in the two groups.
Right ventricular longitudinal strains - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular longitudinal strains in resting conditions using 2D echocardiography in the two groups.
Right ventricular longitudinal strain rates - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular longitudinal strain rates in resting conditions using 2D echocardiography in the two groups.
Left atrial longitudinal strain rates - 2D | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left atrial longitudinal strain rate components in resting conditions using 2D echocardiography in the two groups.
Intraventricular pressure gradient | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess intraventricular pressure gradient of the left ventricle in resting conditions using 2D echocardiography in the two groups.
Vorticity indexes | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular vorticity indexes in resting conditions using 2D echocardiography in the two groups.
Kinetic energy of left ventricular flow | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess kinetic energy of left ventricular flow in resting conditions using 2D echocardiography in the two groups.
Left ventricular wall thicknesses | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular wall thicknesses in resting conditions using echocardiography in the two groups.
Left ventricular diameters | From date of enrollment until the date of evaluation, assessed up to 1 month..
  The investigators will assess left ventricular diameters in resting conditions using echocardiography in the two groups.
Left ventricular volumes | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular volumes in resting conditions using echocardiography in the two groups.
Left ventricular mass | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular mass in resting conditions using echocardiography in the two groups.
Left ventricular ejection fraction | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular ejection fraction in resting conditions using echocardiography in the two groups.
Left ventricular Tissue Doppler Imaging | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular myocardial velocities in resting conditions using echocardiography in the two groups.
Left ventricular transmitral flow | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular transmitral flow in resting conditions using echocardiography in the two groups.
Left ventricular filling pressure index | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left ventricular filling pressure index in resting conditions using echocardiography in the two groups.
Right ventricular outflow tract diameter | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular outflow tract diameter in resting conditions using echocardiography in the two groups.
Tricuspid annular plane systolic excursion | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess tricuspid annular plane systolic excursion in resting conditions using echocardiography in the two groups.
Right ventricular fractional area change | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular fractional area change in resting conditions using echocardiography in the two groups.
Right ventricular ejection fraction | From date of enrollment until the date of evaluation, assessed up to 1 month..
  The investigators will assess right ventricular ejection fraction in resting conditions using echocardiography in the two groups.
Right ventricular Tissue Doppler Imaging | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular myocardial velocities in resting conditions using echocardiography in the two groups.
Right ventricular transtricuspid flow | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular transtricuspid flow in resting conditions using echocardiography in the two groups.
Right ventricular filling pressure gradient | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular filling pressure gradient in resting conditions using echocardiography in the two groups.
Right ventricular systolic pressure | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right ventricular systolic pressure in resting conditions using echocardiography in the two groups.
Left atrial volumes | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess left atrial volumes in resting conditions using echocardiography in the two groups.
Right atrial volumes | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess right atrial volumes in resting conditions using echocardiography in the two groups.
Blood pressures | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess blood pressures in resting conditions using a tensiometer in the two groups.
Heart rate | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess heart rate in resting conditions using echocardiography in the two groups.
Stroke volume | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess stroke volume in resting conditions using echocardiography in the two groups.
Cardiac output | From date of enrollment until the date of evaluation, assessed up to 1 month.
  The investigators will assess cardiac output in resting conditions using echocardiography in the two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - LaPEC, Avignon
  - CHU Montpellier, Montpellier